CLINICAL TRIAL: NCT04702386
Title: Experiences, Expectations and Needs of Children Whose Parents Have Cystic Fibrosis - Exploratory Study
Brief Title: Concerns of Children Whose Parents Have Cystic Fibrosis
Acronym: MUCOKIDS
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Grégory Lemarchal Association (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190326
Record Dates: First submitted 2021-01-07; First posted 2021-01-08 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; parenthood; child with a severely ill parent; Psycho-social; Qualitative study
MeSH Terms: conditions — Cystic Fibrosis | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Focus groups: Children aged 8 years or more participating in a focus group with the study psychologist
  Interventions: Behavioral: Focus groups; Behavioral: Individual interviews
- Individual interviews: All children who have an individual interview with the study psychologist
  Interventions: Behavioral: Focus groups; Behavioral: Individual interviews

INTERVENTIONS:
Behavioral: Focus groups — Groups of 3 to 8 children led by the study psychologist lasting 1 hour for the 8-11-year-old children and up to 2 hours for the children of at least 12 years old, about being the child of a parent with CF
Behavioral: Individual interviews — Interview led by the psychologist about being the child of a parent with CF

SUMMARY:
As more and more patients with cystic fibrosis (CF) become parents, we have studied parenting concerns in this serious chronic disease in a first study (MucoPar) which is ongoing.

The current study (MucoKids) is an extension of the previous MucoPar study and aims to explore and collect the perceptions, expectations and needs of children whose one parent has CF.

This will be done in the context of individual interviews or in several small groups of children led by a psychologist who will encourage them to develop what constitutes to be the child of somebody with CF.

The collected information should make it possible to develop and propose adapted medico-psycho-social interventions, if necessary, in connection with patient associations.

DETAILED DESCRIPTION:
Life expectancy has improved significantly in cystic fibrosis in recent years. From pediatric disease, it has become a disease of the adult, with the emergence of new issues, such as becoming a parent. Parent patients still face the risk of complications and death while their child is still young. However, there is very little data in the literature on parenting in cystic fibrosis. In a first study which is ongoing (43 patients out of the 50 planned have been included), we intended to study parenting, considering the sick parent's point of view.

However, this question does not only concern parents and their spouses. It is also fundamental to take into account the experience of the children, to understand their experiences and their own needs in this context of serious illness of a parent with limited life expectancy.

Therefore, the purpose of this study is to explore and collect the perceptions, expectations and needs of children whose one parent has CF. Children are eligible from the age of 6 if their parents agree.

Children will have semi-structured individual interviews or will participate in focus groups with the study psychologist in order to express their feelings, difficulties, expectations and needs in living with a parent who has CF.

Thematic analysis of the content will first be done separately for individual interviews and focus groups, and a global synthesis will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Have a parent with CF cared at one of the 2 adult CF centres participating into the study
* Have the authorization of the parent with CF if the child is an adult and of both parents for subjects less than 18 years old
* Be ay least 6 years old
* Have a good level of French and good speaking skills for adolescents and adults
* Have a level of French and oral expression skills adapted to their age group for the youngest

Exclusion Criteria:

* Psychiatric pathology (borderline state, bipolarity and other psychotic disorders) in their parents or themselves
* Serious somatic disease not related to cystic fibrosis in their parents or themselves

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is comprised of people, both minors and adults, who have a parent living with cystic fibrosis. These parents are participants in the study MUCOPAR.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Identification of themes about being the child of a parent with CF | 2 years
  Content of groups and individual interviews analysed by thematic analysis

SECONDARY OUTCOMES:
Occurrence of themes | 2 years
  The number of appearances of each theme, in focus groups and in individual interviews will provide information on the importance of each theme.

CONTACTS AND LOCATIONS:
Overall Officials: Cécile FLAHAULT, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris; Dominique HUBERT, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Cochin Hospital, Paris
  - Foch Hospital, Suresnes

IPD SHARING:
Plan to Share IPD: No